CLINICAL TRIAL: NCT00889798
Title: Epidemiological Registry Describing Treatment Reality and Therapy Modalities of Patients With Malignant Lymphatic Systemic Diseases (Non-Hodgkin's Lymphoma, Chronic Lymphocytic Leukemia and Multiple Myeloma) Requiring Therapy.
Brief Title: Tumor Registry of Lymphatic Neoplasia
Acronym: TLN-Registry
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-TLN
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Non-Hodgkin's Lymphoma (NHL); Chronic Lymphocytic Leukemia (CLL); Multiple Myeloma (MM)
Keywords: Malignant lymphatic disease; therapy-reality; observation; registry; therapy sequences; NHL; CLL; Germany; lenalidomide; alemtuzumab; rituximab; bendamustin; thalidomide; bortezomib; ibritumomab-tiuxetan; G-CSF (Granulocyte-Colony Stimulating Factor); chronic lymphocytic leukaemia; follicular lymphoma; gastric MALT lymphoma (Mucosa Associated Lymphoid Tissue); nongastric MALT lymphoma (Mucosa Associated Lymphoid Tissue); nodal marginal zone lymphoma; splenic marginal zone lymphoma; mantle cell lymphoma; diffuse large b-cell lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Leukemia, B-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this registry is to record information on therapy reality of malignant lymphatic systemic diseases by office-based haematologists in Germany.

DETAILED DESCRIPTION:
The TLN is a prospective, longitudinal, nation wide cohort study with the purpose to record information on the antineoplastic treatment of lymphatic neoplasms in Germany. The registry will follow patients for up to five years. It will identify common therapeutic sequences and changes in the treatment of the disease. At inclusion, data in patient characteristics, comorbidities, tumor characteristics and previous treatments are collected. During the course of observation data on all systemic treatments, radiotherapies, surgeries, and outcome are documented.

The impact of nutrition (LyNut) and physical activity (LyNut) on the course of the adjuvant disease will be examined in patients with indolent and aggressive Non-Hodgin Lymphoma, as well as long-term effects of systemic treatment (LyTox) and quality of life (LyLife) in patients with multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Non-Hodgkin's lymphoma, chronic lymphocytic leukaemia or multiple myeloma
* Must receive a first- or second-line therapy
* 18 years or older
* Signed, written informed consent

Exclusion Criteria:

- no systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a malignant lymphatic disease requiring therapy
Sampling Method: Non-Probability Sample
Enrollment: 3795 (Actual)
Dates: Start 2009-04; Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Course of treatment (treatment reality) | 5 years per patient
  Documentation of anamnestic data and therapy sequences

SECONDARY OUTCOMES:
Effectiveness of treatment | 5 years per patient
  Documentation of response rates and progression-free survival per therapy sequence, overall survival time and adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Knauf, MD, Study Chair — Center for Haematology, Frankfurt, Germany; Wolfang Abenhardt, MD, Study Chair — MVZ Onkologie im Elisenhof, München, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Knauf W, Abenhardt W, Dorfel S, Meyer D, Grugel R, Munz M, Hartmann H, Marschner N. Routine treatment of patients with chronic lymphocytic leukaemia by office-based haematologists in Germany-data from the Prospective Tumour Registry Lymphatic Neoplasms. Hematol Oncol. 2015 Mar;33(1):15-22. doi: 10.1002/hon.2139. Epub 2014 Apr 15. PMID 24733536
- [Result] Knauf W, Abenhardt W, Aldaoud A, Nusch A, Grugel R, Munz M, Hartmann H, Marschner N; TLN Study Group. Treatment of Non-transplant patients with multiple myeloma: routine treatment by office-based haematologists in Germany--data from the prospective Tumour Registry Lymphatic Neoplasms (TLN). Oncol Res Treat. 2014;37(11):635-6, 638-44. doi: 10.1159/000368315. Epub 2014 Oct 17. PMID 25486127
- [Result] Knauf W, Aldaoud A, Hutzschenreuter U, Klausmann M, Dille S, Wetzel N, Janicke M, Marschner N; and the TLN-Group (Tumour Registry Lymphatic Neoplasms). Survival of non-transplant patients with multiple myeloma in routine care differs from that in clinical trials-data from the prospective German Tumour Registry Lymphatic Neoplasms. Ann Hematol. 2018 Dec;97(12):2437-2445. doi: 10.1007/s00277-018-3449-8. Epub 2018 Aug 1. PMID 30069704
- [Result] Knauf W, Abenhardt W, Mohm J, Rauh J, Harde J, Kaiser-Osterhues A, Janicke M, Marschner N; TLN-Group (Tumour Registry Lymphatic Neoplasms). Similar effectiveness of R-CHOP-14 and -21 in diffuse large B-cell lymphoma-data from the prospective German Tumour Registry Lymphatic Neoplasms. Eur J Haematol. 2019 Nov;103(5):460-471. doi: 10.1111/ejh.13295. Epub 2019 Sep 4. PMID 31314918
- [Result] Knauf W, Abenhardt W, Slawik HR, Buckner U, Otremba B, Sauer A, Zahn MO, Wetzel N, Kaiser-Osterhues A, Houet L, Marschner N; TLN-Group (Tumour Registry Lymphatic Neoplasms). Rare lymphomas in routine practice-Treatment and outcome in Waldenstrom's macroglobulinaemia in the prospective German Tumour Registry Lymphatic Neoplasms. Hematol Oncol. 2020 Aug;38(3):344-352. doi: 10.1002/hon.2740. Epub 2020 May 8. PMID 32383192